CLINICAL TRIAL: NCT02028754
Title: A Study of Sodium Carboxymethylcellulose for Post Cataract Surgery Dry Eye Symptoms
Acronym: RLOTUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN-CMC-1101
Record Dates: First submitted 2014-01-06; First posted 2014-01-07 (Estimated); Results first posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-03

CONDITIONS: Dry Eye Syndromes; Cataract
MeSH Terms: conditions — Dry Eye Syndromes; Cataract | interventions — Carboxymethylcellulose Sodium; Levofloxacin; Prednisolone; prednisolone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium Carboxymethylcellulose and Conventional Therapy (Experimental): Sodium carboxymethylcellulose (Refresh Liquigel®) 1 drop in the study eye 4 times a day for 30 days plus conventional therapy of levofloxacin for 7 days post-cataract surgery and prednisolone for 30 days post-cataract surgery each in the study eye up to 4 times a day.
  Interventions: Drug: Sodium Carboxymethylcellulose; Drug: Levofloxacin; Drug: Prednisolone
- Conventional Therapy (Active Comparator): Conventional therapy of levofloxacin for 7 days post-cataract surgery and prednisolone for 30 days post-cataract surgery each in the study eye up to 4 times a day.
  Interventions: Drug: Levofloxacin; Drug: Prednisolone

INTERVENTIONS:
Drug: Sodium Carboxymethylcellulose — Sodium carboxymethylcellulose (Refresh Liquigel®) 1 drop in the study eye 4 times a day for 30 days post-cataract surgery.
  Other Names: Refresh Liquigel®
  Arms: Sodium Carboxymethylcellulose and Conventional Therapy
Drug: Levofloxacin — Levofloxacin 1 drop in the study eye 3 times a day for 7 days post-cataract surgery.
  Other Names: Cravit®
Drug: Prednisolone — Prednisolone 1 drop in the study eye 4 times a day for the 1st week post surgery, 3 times a day for the 2nd week post surgery, 2 times a day for the 3rd week post surgery, and 1 time a day for the 4th week post surgery.
  Other Names: PRED FORTE®

SUMMARY:
This study will evaluate the effect of sodium carboxymethylcellulose eye drops in the treatment of dry eye after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of age-related cataract in the study eye
* Scheduled for cataract surgery and lens implant

Exclusion Criteria:

* Diagnosis of ocular surface disease or glaucoma
* Ocular surgery in the past 3 months
* Wearing a corneal contact lens in the study eye

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2011-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Hangzhou, China

REFERENCES:
- [Derived] Yao K, Bao Y, Ye J, Lu Y, Bi H, Tang X, Zhao Y, Zhang J, Yang J. Efficacy of 1% carboxymethylcellulose sodium for treating dry eye after phacoemulsification: results from a multicenter, open-label, randomized, controlled study. BMC Ophthalmol. 2015 Mar 20;15:28. doi: 10.1186/s12886-015-0005-3. PMID 25880685

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sodium Carboxymethylcellulose and Conventional Therapy | Conventional Therapy
Started | 90 | 90
Completed | 83 | 82
Not Completed | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Carboxymethylcellulose and Conventional Therapy | Conventional Therapy | Total
Number analyzed (Participants) | 90 | 90 | 180
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.8 (7.1) | 69.0 (7.1) | 68.9 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 59 | 113
  Male | 36 | 31 | 67

OUTCOME MEASURES:

1. Primary Outcome: Tear Break-Up Time (TBUT) in the Study Eye
Description: TBUT is the time required for dry spots to appear on the surface of the study eye after blinking. The longer it takes, the more stable the tear film. A short TBUT is a sign of poor tear film.
Time Frame: Day 7
Population: All patients with data at this time point
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Sodium Carboxymethylcellulose and Conventional Therapy | Conventional Therapy
Number analyzed (Participants) | 85 | 85
Seconds | 8.5 (5.5) | 6.6 (3.8)

2. Primary Outcome: Tear Break-Up Time (TBUT) in the Study Eye
Description: as for outcome 1
Time Frame: Day 30
Population: All patients with data at this time point
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Sodium Carboxymethylcellulose and Conventional Therapy | Conventional Therapy
Number analyzed (Participants) | 83 | 82
Seconds | 9.0 (5.9) | 6.7 (4.8)

3. Secondary Outcome: Fluorescein Staining Score in the Study Eye
Description: The cornea is evaluated following ocular administration of fluorescein stain in the study eye. The cornea is the transparent front part of the eye which covers the iris and pupil. The cornea is divided into 3 regions. Each region is scored according to the extent of staining, with scores ranging from 0 to 3 points: 0=non-staining, 1=staining range < 1/2 of the cornea, 2=staining range ≥ 1/2 of the cornea, and 3=regional whole staining of the cornea. The total score ranges from 0 to 9 points. The higher the staining score, the worse the dry eye condition.
Time Frame: Day 7, Day 30
Population: All patients with data at this time point
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Sodium Carboxymethylcellulose and Conventional Therapy | Conventional Therapy
Number analyzed (Participants) | 85 | 85
Scores on a Scale
  Day 7 | 2.0 (2.8) | 1.8 (2.6)
  Day 30 (N=83, 82) | 1.1 (1.8) | 1.2 (1.9)

4. Secondary Outcome: Lissamine Green Staining Score in the Study Eye
Description: Conjunctival and corneal staining are evaluated following ocular administration of lissamine green dye in the study eye. The conjunctiva is the clear membrane covering the white surface of the eye. The cornea is the transparent front part of the eye which covers the iris and pupil. The conjunctiva and cornea are divided into 5 regions that are scored based on the extent of staining. Scores range from 0 to 3 points: 0=non-staining, 1=staining range < 1/2 of the conjunctiva and cornea, 2=staining range ≥ 1/2 of the conjunctiva and cornea, and 3=regional whole staining of the conjunctiva and cornea. The total score ranges from 0 to 15 points. The higher the grade score, the worse the dry eye condition.
Time Frame: Day 7, Day 30
Population: All patients with data at this time point
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Sodium Carboxymethylcellulose and Conventional Therapy | Conventional Therapy
Number analyzed (Participants) | 85 | 85
Scores on a Scale
  Day 7 | 2.9 (3.3) | 2.6 (3.2)
  Day 30 (N=83,82) | 2.1 (2.4) | 2.3 (2.6)

5. Secondary Outcome: Results of Schirmer I Test With Anesthetics in the Study Eye
Description: The Schirmer I test consists of anesthetic drops being placed into the lower eyelid of the study eye. Patients then close their eyes. Test paper is placed on the lower eyelid of the patient's closed eyes. The paper is then removed and the moisture length on the paper recorded. Shorter distances indicate worse dry eye symptoms.
Time Frame: Day 7, Day 30
Population: All patients with data at this time point
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Sodium Carboxymethylcellulose and Conventional Therapy | Conventional Therapy
Number analyzed (Participants) | 85 | 85
Millimeters
  Day 7 | 11.8 (5.6) | 12.5 (6.8)
  Day 30 (N=83, 82) | 12.7 (6.1) | 12.6 (6.5)

6. Secondary Outcome: Ocular Surface Disease Index (OSDI) Questionnaire Score in the Study Eye
Description: The OSDI is a 12-question survey for patients to document their dry eye disease symptoms in the study eye. The OSDI consists of a 5-point scale (0=none of the time and 4 = all of the time), with higher scores representing greater disability. The scores are totaled over the 12 questions and converted to a score of 0-100 (0=no disability and 100=complete disability).
Time Frame: Day 7, Day 30
Population: All patients with data at this time point
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Sodium Carboxymethylcellulose and Conventional Therapy | Conventional Therapy
Number analyzed (Participants) | 85 | 85
Scores on a Scale
  Day 7 | 15.6 (16.8) | 18.1 (19.5)
  Day 30 (N=83, 82) | 12.7 (11.3) | 14.2 (13.8)

7. Secondary Outcome: Subjective Symptom Total Score in the Study Eye
Description: The following 11 subjective symptoms are evaluated in the study eye: foreign body sensation, photophobia, itching, pain in the eye, dry eye, eye heaviness, blurred vision, eye fatigue, eye discomfort, eye secretions and tears. Each of these symptoms is divided into 4 classes: no symptom=0; occasional symptoms=1; intermittent mild symptoms=2; and persistent obvious symptoms=3. The total score ranged from 0 (best) to 33 (worst).
Time Frame: Day 7, Day 30
Population: All patients with data at this time point
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Sodium Carboxymethylcellulose and Conventional Therapy | Conventional Therapy
Number analyzed (Participants) | 85 | 85
Scores on a Scale
  Day 7 | 6.1 (5.3) | 6.4 (5.2)
  Day 30 (N=83, 82) | 5.1 (3.6) | 5.6 (4.0)

ADVERSE EVENTS:
Description: The Safety Population included all patients with safety data and was used to evaluate adverse events (AEs) and serious adverse events (SAEs).
Arm/Group | Sodium Carboxymethylcellulose and Conventional Therapy | Conventional Therapy
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/85
Other Adverse Events (participants affected / at risk) | 0/86 | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is at least 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.